CLINICAL TRIAL: NCT05941624
Title: Comparison Between HA330 Hemoperfusion Filter Hemodialysis and Conventional High-Flux Filter Hemodialysis in Reducing Inflammatory Mediators in Renal Dysfunction Due to Sepsis
Brief Title: Comparison Between HA330 Hemoperfusion Filter Hemodialysis and Conventional High-Flux Hemodialysis Filter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, Principal investigator, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IndonesiaUAnes043
Record Dates: First submitted 2023-06-20; First posted 2023-07-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Renal Dysfunction; Sepsis; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ha-330 Hemoperfusion Filter Hemodialysis (Experimental): Participants underwent therapy using Ha-330 Hemoperfusion Filter Hemodialysis for 4 hours, 3 times a week, with two days apart between dialysis.
  Interventions: Device: Ha-330 Hemoperfusion Filter Hemodialysis
- Conventional hemodialysis (Active Comparator): Participants underwent therapy using Conventional Hemodialysis for 4 hours, 3 times a week, with two days apart between dialysis.
  Interventions: Device: Conventional Hemodialysis

INTERVENTIONS:
Device: Ha-330 Hemoperfusion Filter Hemodialysis — a total of 4 hours therapy, 3 times a week. Each therapy should be two days apart
  Arms: Ha-330 Hemoperfusion Filter Hemodialysis
Device: Conventional Hemodialysis — a total of 4 hours therapy, 3 times a week. Each therapy should be two days apart
  Arms: Conventional hemodialysis

SUMMARY:
The purpose of this study is to compare the effectiveness between conventional hemodialysis and hemodialysis using hemoperfusion adsorbents in renal dysfunction caused by sepsis

DETAILED DESCRIPTION:
This study is an open randomized clinical trial. Data were taken prospectively until the number of samples was fulfilled for analysis. Due to the intervention provided, this study was not blinded. Subjects were divided into 2 groups (group undergoing conventional hemodialysis and group undergoing HA330 hemoperfusion). Both groups underwent therapy for 4 hours, 3 times a week, with two days apart between dialysis. Inflammatory mediator levels were assessed 4 times, before and after each intervention. All subjects were given standard therapy as indicated such as antibiotics, oxygen supplementation, administration of vasopressors, nutrition, and other therapies as indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 - 65 years old
* Patients diagnosed with sepsis with acute kidney injury whose indicated for hemodialysis. Including fluid overload, life-threatening metabolic acidosis, hypercalcemia, pulmonary edema, and uremic

Exclusion Criteria:

* Patients with hemodynamic instability who need norepinephrine more than 0.5 microgram/kg/minute
* Patients denied to be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Interleukin (IL)-1Ra concentration before and after hemodialysis | 1 week
  IL-1Ra measurement using ELISA from 5 mL of veins from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. IL-1Ra will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Change in Interleukin (IL)-6 concentration before and after hemodialysis | 1 week
  IL-6 measurement using ELISA from 5 mL of veins from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. IL-6 will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Change in Interleukin (IL)-10 concentration before and after hemodialysis | 1 week
  IL-10 measurement using ELISA from 5 mL of veins from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. IL-10 will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Change in Tumor Necrosis Factor (TNF)-a concentration before and after hemodialysis | 1 week
  TNF-a measurement using ELISA from 5 mL of veins from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. TNF-a will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.

SECONDARY OUTCOMES:
Leukocytes Levels | 1 week
  Leukocytes measurement using automatic hematology analyzer. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Leukocytes will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Neutrophils Levels | 1 week
  Neutrophil measurement using automatic hematology analyzer. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Neutrophils will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Lymphocytes Levels | 1 week
  Lymphocytes measurement using automatic hematology analyzer. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Lymphocytes will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Thrombocytes Levels | 1 week
  Thrombocytes measurement using automatic hematology analyzer. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Lymphocytes will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
C-Reactive Protein (CRP) Levels | 1 week
  C-Reactive Protein measurement using latex agglutination method. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. CRP levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Procalcitonin Levels | 1 week
  Procalcitonin measurement using particle enhanced immunoturbidimetric test. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Procalcitonin levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Urea Levels | 1 week
  Urea measurement using enzymatic method (Glutamate dehydrogenase). The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Urea levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Creatinine Levels | 1 week
  Creatinine measurement using Calorimetry. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Creatinine levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Glomerular Filtration Rate (GFR) | 1 week
  Glomerular Filtration Rate measurement with creatinine clearance test using the Cockcroft-Gault formula
Bilirubin Levels | 1 week
  Total bilirubin measurement with DCA method (Colorimetry test-Dichloroaniline). The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Bilirubin levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Serum Glutamic Oxaloacetic Transaminase (SGOT) Levels | 1 week
  Serum glutamic oxaloacetic transaminase measurement with kinetic method using spectrophotometer. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. SGOT will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Serum Glutamic Pyruvate Transaminase (SGPT) Levels | 1 week
  Serum glutamic pyruvate transaminase measurement with kinetic method using spectrophotometer. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. SGPT will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Prothrombin Time (PT) | 1 week
  Prothrombin time measurement using optical/mechanical photo. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. PT levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Activated Partial Thromboplastin Time (aPTT) | 1 week
  Activated partial thromboplastin Time measurement using optical/mechanical photo. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. aPTT levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
International Normalizing Ratio (INR) | 1 week
  International normalizing ratio measurement using optical/mechanical photo. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. INR will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Lactate Levels | 1 week
  Lactate measurement using lactate oxidase. The sample is taken from 5 mL of venous blood from central venous catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Lactate levels will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Blood pH (Potential Hydrogen) | 1 week
  Blood pH measurement using the pH indicator into blood sample for some minutes. The sample is taken from 3 mL of arterial blood from arterial catheter from baseline (1 hour before first intervention) and 1 hour after intervention. SGPT will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Base Excess (BE) | 1 week
  Base Excess measurement using 2 methods: direct and blood gas analysis. The sample is taken from 3 mL of arterial blood from arterial catheter from baseline (1 hour before first intervention) and 1 hour after intervention. Base excess will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
PaO2 (Partial pressure of oxygen) | 1 week
  PaO2 measurement using gasometry and osmometry methods. The sample is taken from 3 mL of arterial blood from arterial catheter from baseline (1 hour before first intervention) and 1 hour after intervention. PaO2 will also be measured at the 2nd (day 3) and 3rd (day 5) therapy, 1 hour before and 1 hour after treatment each.
Mean Arterial Pressure (MAP) | 1 week
  Mean Arterial Pressure is calculated using the MAP formula (Systole + 2 x diastole) / 3
Heart Rate | 1 week
  Heart rate measured manually from the left radial artery for 1 minute
Vasoactive Drugs needed | 1 week
  Highest dosage of vasoactive drugs during the intervention
Mortality | 30 days
  Data extracted from medical record
Length of Stay in ICU | 30 days
  Length of ICU stay in days from admission until the patient meets the ICU discharge criteria
Length of Stay in Hospital | 30 days
  Length of hospital stay in days from admission until the patient discharged from the hospital
Post ICU Routine Hemodialysis Need | 30 days
  Data extracted from medical record
Fluid Status | 1 - 2 week
  Fluid Status was measured using Bioelectrical Impedance Analysis. The fluid status is represented from Extracellular Water (ECW), Intracellular Water (ICW), and Total Body Water (TBW). Measurements are conducted 1 hour Pre and Post Hemodialysis 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Dita Aditianingsih, M.D., Principal Investigator — Indonesia University
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Susantitaphong P, Cruz DN, Cerda J, Abulfaraj M, Alqahtani F, Koulouridis I, Jaber BL; Acute Kidney Injury Advisory Group of the American Society of Nephrology. World incidence of AKI: a meta-analysis. Clin J Am Soc Nephrol. 2013 Sep;8(9):1482-93. doi: 10.2215/CJN.00710113. Epub 2013 Jun 6. PMID 23744003
- [Background] Uchino S, Kellum JA, Bellomo R, Doig GS, Morimatsu H, Morgera S, Schetz M, Tan I, Bouman C, Macedo E, Gibney N, Tolwani A, Ronco C; Beginning and Ending Supportive Therapy for the Kidney (BEST Kidney) Investigators. Acute renal failure in critically ill patients: a multinational, multicenter study. JAMA. 2005 Aug 17;294(7):813-8. doi: 10.1001/jama.294.7.813. PMID 16106006
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Ronco C, Ricci Z, De Backer D, Kellum JA, Taccone FS, Joannidis M, Pickkers P, Cantaluppi V, Turani F, Saudan P, Bellomo R, Joannes-Boyau O, Antonelli M, Payen D, Prowle JR, Vincent JL. Renal replacement therapy in acute kidney injury: controversy and consensus. Crit Care. 2015 Apr 6;19(1):146. doi: 10.1186/s13054-015-0850-8. PMID 25887923
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Ahmed AR, Obilana A, Lappin D. Renal Replacement Therapy in the Critical Care Setting. Crit Care Res Pract. 2019 Jul 16;2019:6948710. doi: 10.1155/2019/6948710. eCollection 2019. PMID 31396416
- [Background] Ankawi G, Fan W, Pomare Montin D, Lorenzin A, Neri M, Caprara C, de Cal M, Ronco C. A New Series of Sorbent Devices for Multiple Clinical Purposes: Current Evidence and Future Directions. Blood Purif. 2019;47(1-3):94-100. doi: 10.1159/000493523. Epub 2018 Sep 25. PMID 30253409
- [Background] Rudd KE, Johnson SC, Agesa KM, Shackelford KA, Tsoi D, Kievlan DR, Colombara DV, Ikuta KS, Kissoon N, Finfer S, Fleischmann-Struzek C, Machado FR, Reinhart KK, Rowan K, Seymour CW, Watson RS, West TE, Marinho F, Hay SI, Lozano R, Lopez AD, Angus DC, Murray CJL, Naghavi M. Global, regional, and national sepsis incidence and mortality, 1990-2017: analysis for the Global Burden of Disease Study. Lancet. 2020 Jan 18;395(10219):200-211. doi: 10.1016/S0140-6736(19)32989-7. PMID 31954465
- [Background] Chousterman BG, Swirski FK, Weber GF. Cytokine storm and sepsis disease pathogenesis. Semin Immunopathol. 2017 Jul;39(5):517-528. doi: 10.1007/s00281-017-0639-8. Epub 2017 May 29. PMID 28555385
- [Background] Murugan R, Karajala-Subramanyam V, Lee M, Yende S, Kong L, Carter M, Angus DC, Kellum JA; Genetic and Inflammatory Markers of Sepsis (GenIMS) Investigators. Acute kidney injury in non-severe pneumonia is associated with an increased immune response and lower survival. Kidney Int. 2010 Mar;77(6):527-35. doi: 10.1038/ki.2009.502. Epub 2009 Dec 23. PMID 20032961
- [Background] Fiorentino M, Tohme FA, Wang S, Murugan R, Angus DC, Kellum JA. Long-term survival in patients with septic acute kidney injury is strongly influenced by renal recovery. PLoS One. 2018 Jun 5;13(6):e0198269. doi: 10.1371/journal.pone.0198269. eCollection 2018. PMID 29870535
- [Background] Alobaidi R, Basu RK, Goldstein SL, Bagshaw SM. Sepsis-associated acute kidney injury. Semin Nephrol. 2015 Jan;35(1):2-11. doi: 10.1016/j.semnephrol.2015.01.002. PMID 25795495
- [Background] Schneider AG, Bellomo R, Bagshaw SM, Glassford NJ, Lo S, Jun M, Cass A, Gallagher M. Choice of renal replacement therapy modality and dialysis dependence after acute kidney injury: a systematic review and meta-analysis. Intensive Care Med. 2013 Jun;39(6):987-97. doi: 10.1007/s00134-013-2864-5. Epub 2013 Feb 27. PMID 23443311
- [Background] Sood MM, Shafer LA, Ho J, Reslerova M, Martinka G, Keenan S, Dial S, Wood G, Rigatto C, Kumar A; Cooperative Antimicrobial Therapy in Septic Shock (CATSS) Database Research Group. Early reversible acute kidney injury is associated with improved survival in septic shock. J Crit Care. 2014 Oct;29(5):711-7. doi: 10.1016/j.jcrc.2014.04.003. Epub 2014 Apr 18. PMID 24927984
- [Background] See EJ, Jayasinghe K, Glassford N, Bailey M, Johnson DW, Polkinghorne KR, Toussaint ND, Bellomo R. Long-term risk of adverse outcomes after acute kidney injury: a systematic review and meta-analysis of cohort studies using consensus definitions of exposure. Kidney Int. 2019 Jan;95(1):160-172. doi: 10.1016/j.kint.2018.08.036. Epub 2018 Nov 23. PMID 30473140
- [Background] Chawla LS, Amdur RL, Amodeo S, Kimmel PL, Palant CE. The severity of acute kidney injury predicts progression to chronic kidney disease. Kidney Int. 2011 Jun;79(12):1361-9. doi: 10.1038/ki.2011.42. Epub 2011 Mar 23. PMID 21430640
- [Background] Chua HR, Wong WK, Ong VH, Agrawal D, Vathsala A, Tay HM, Mukhopadhyay A. Extended Mortality and Chronic Kidney Disease After Septic Acute Kidney Injury. J Intensive Care Med. 2020 Jun;35(6):527-535. doi: 10.1177/0885066618764617. Epub 2018 Mar 18. PMID 29552953
- [Background] Zarjou A, Agarwal A. Sepsis and acute kidney injury. J Am Soc Nephrol. 2011 Jun;22(6):999-1006. doi: 10.1681/ASN.2010050484. Epub 2011 May 12. PMID 21566052
- [Background] Peerapornratana S, Manrique-Caballero CL, Gomez H, Kellum JA. Acute kidney injury from sepsis: current concepts, epidemiology, pathophysiology, prevention and treatment. Kidney Int. 2019 Nov;96(5):1083-1099. doi: 10.1016/j.kint.2019.05.026. Epub 2019 Jun 7. PMID 31443997
- [Background] Megha KB, Joseph X, Akhil V, Mohanan PV. Cascade of immune mechanism and consequences of inflammatory disorders. Phytomedicine. 2021 Oct;91:153712. doi: 10.1016/j.phymed.2021.153712. Epub 2021 Aug 19. PMID 34511264
- [Background] Mishra SB, Singh RK, Baronia AK, Poddar B, Azim A, Gurjar M. Sustained low-efficiency dialysis in septic shock: Hemodynamic tolerability and efficacy. Indian J Crit Care Med. 2016 Dec;20(12):701-707. doi: 10.4103/0972-5229.195704. PMID 28149027
- [Background] Huang Z, Wang SR, Su W, Liu JY. Removal of humoral mediators and the effect on the survival of septic patients by hemoperfusion with neutral microporous resin column. Ther Apher Dial. 2010 Dec;14(6):596-602. doi: 10.1111/j.1744-9987.2010.00825.x. PMID 21118369
- [Background] Bagshaw SM, Berthiaume LR, Delaney A, Bellomo R. Continuous versus intermittent renal replacement therapy for critically ill patients with acute kidney injury: a meta-analysis. Crit Care Med. 2008 Feb;36(2):610-7. doi: 10.1097/01.CCM.0B013E3181611F552. PMID 18216610
- [Background] Hu XB, Gao HB, Liao ME, He MR. [The use of HA330-II microporous resin plasma adsorption in the treatment of chronic severe hepatitis]. Zhongguo Wei Zhong Bing Ji Jiu Yi Xue. 2007 Dec;19(12):760-1. No abstract available. Chinese. PMID 18093442
- [Background] Sun S, He L, Bai M, Liu H, Li Y, Li L, Yu Y, Shou M, Jing R, Zhao L, Huang C, Wang H. High-volume hemofiltration plus hemoperfusion for hyperlipidemic severe acute pancreatitis: a controlled pilot study. Ann Saudi Med. 2015 Sep-Oct;35(5):352-8. doi: 10.5144/0256-4947.2015.352. PMID 26506968
- [Background] Bai M, Yu Y, Huang C, Liu Y, Zhou M, Li Y, Ma F, Jing R, Zhao L, Li L, Wang P, He L, Sun S. Continuous venovenous hemofiltration combined with hemoperfusion for toxic epidermal necrolysis: a retrospective cohort study. J Dermatolog Treat. 2017 Jun;28(4):353-359. doi: 10.1080/09546634.2016.1240326. Epub 2016 Oct 24. PMID 27653468
- [Background] Kacar CK, Uzundere O, Kandemir D, Yektas A. Efficacy of HA330 Hemoperfusion Adsorbent in Patients Followed in the Intensive Care Unit for Septic Shock and Acute Kidney Injury and Treated with Continuous Venovenous Hemodiafiltration as Renal Replacement Therapy. Blood Purif. 2020;49(4):448-456. doi: 10.1159/000505565. Epub 2020 Jan 28. PMID 31991412
- [Background] Li J, Li H, Deng W, Meng L, Gong W, Yao H. The Effect of Combination Use of Hemodialysis and Hemoperfusion on Microinflammation in Elderly Patients with Maintenance Hemodialysis. Blood Purif. 2022;51(9):739-746. doi: 10.1159/000518857. Epub 2022 Jan 14. PMID 36096108
- [Background] Coudroy R, Payen D, Launey Y, Lukaszewicz AC, Kaaki M, Veber B, Collange O, Dewitte A, Martin-Lefevre L, Jabaudon M, Kerforne T, Ferrandiere M, Kipnis E, Vela C, Chevalier S, Mallat J, Charreau S, Lecron JC, Robert R; ABDOMIX group. Modulation by Polymyxin-B Hemoperfusion of Inflammatory Response Related to Severe Peritonitis. Shock. 2017 Jan;47(1):93-99. doi: 10.1097/SHK.0000000000000725. PMID 27984535